CLINICAL TRIAL: NCT03421574
Title: Phase I Trial of MR-guided Focused Ultrasound (MRgFUS) Bilateral Capsulotomy for the Treatment of Refractory Major Depression
Brief Title: Trial of MR-guided Focused Ultrasound for Treatment of Refractory Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Princiapl Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 344-2017
Record Dates: First submitted 2018-01-08; First posted 2018-02-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-Guided Focused Ultrasound (Experimental)
  Interventions: Device: MR-guided Focused Ultrasound

INTERVENTIONS:
Device: MR-guided Focused Ultrasound — Focused Ultrasound allows for non-invasive thermal ablation of soft tissue virtually anywhere in the body. Treatment begins by acquiring a series of magnetic resonance (MR) images of the target tissue. The physician then reviews the images on the system workstation, identifies the target, delineates treatment contours, and reviews the treatment plan. Therapy planning software calculates the parameters required to effectively treat (e.g. ablate) the defined region. During treatment, the patient wears a helmet equipped with multiple sources of ultrasound which generate a point of focused energy, called a sonication. The sonication raises the tissue temperature within a well-defined region, causing a thermal coagulation effect.

SUMMARY:
The proposed study is to evaluate the safety and initial efficacy of MRgFUS for patients with treatment-refractory Major Depression. This study is designed as a prospective, single arm, nonrandomized study. Assessments will be made before and after MRgFUS for adverse events related to treatment, for clinical symptom relief, and quality of life (QoL). The target in the brain chosen for ablation will be the anterior limb of the internal capsule (i.e 'capsulotomy').

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥20 and ≤80 years of age.
2. Patients who are able and willing to give consent and physically and practically able to attend study visits, as determined by both study Psychiatrist and the surgeon.
3. DSM-V diagnosis of major depressive episode, as a component of an Axis I disorder, such as Major Depressive Disorder, Bipolar Disorder, Anxiety Disorder, Eating Disorder, Substance Abuse/Dependence Disorder ,or Personality Disorder
4. At least 5-year illness history of the primary disorder and at least 6 months since the onset of the first episode of major depression.
5. A minimum score of 20 on the Hamilton Depression Rating Scale (HAMD) when depressed (patients with bipolar disorder may be rapid cycling, but have to have at least 2 weeks of major depression at the time the HAMD is conducted)
6. Medication-refractoriness as determined by an adequate dose and duration of standard psychiatric treatments (including psychotherapy and/or pharmacology) as determined by two psychiatrists associated with the study. Including specifically:

   1. Failed to respond or tolerate adequate trial of three or more medications accepted as first line in the treatment of depression
   2. Failed to respond or tolerate augmentation with or combination,of at least 2 medications known to be first line treatments for depression
   3. An adequate trial of cognitive behavioural therapy or other evidence-supported psychotherapy, delivered by a therapist experienced in treating depression
7. Able to communicate sensations during the ExAblate MRgFUS treatment
8. A consistent dose of any and all medications in the 30 days prior to study entry.
9. Women of childbearing potential must agree to use a contraception method throughout the study.

Exclusion Criteria:

1. Patients with unstable cardiac status [e.g. Unstable angina pectoris on medication, Patients with documented myocardial infarction within six months, Congestive heart failure requiring medication (other than diuretic), Patients on anti-arrhythmic drugs, Severe hypertension (diastolic BP > 100 on medication)]
2. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
3. Severely impaired renal function (estimated glomerular filtration rate < 30ml/min/1.73 m2) or receiving dialysis
4. Laboratory biochemical evidence of abnormal bleeding and/or coagulopathy, including risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter or abnormal INR)
5. Cerebrovascular disease (e.g. CVA within 6 months) or history of intracranial hemorrhage
6. Untreated, uncontrolled sleep apnea
7. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
8. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
9. Are participating or have participated in another clinical trial in the last 30 days
10. Patients unable to communicate with the investigator and staff.
11. Presence of significant cognitive impairment
12. Presence of psychosis on clinical evaluation.
13. Patients with brain tumors already known or revealed on pretreatment MRI
14. Currently pregnant (as determined by history and serum HCG) or lactating.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 year
  Safety of the ExAblate transcranial treatment will be determined by an evaluation of the incidence and severity of procedure related complications from the treatment day visit through the 12-month post-treatment time point. All events that are not procedure related will also be captured and recorded.

SECONDARY OUTCOMES:
Quality of Life will be measured using the Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ) | 1 year
  Q-LES-Q) is a self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. The minimum raw score on the Q-LES-Q-SF is 14, and the maximum score is 70.
Clinical efficacy will be measured using the Hamilton Rating Scale for Depression (HAMD) | 1 year
  The HAMD is designed to rate the severity of depression in patients. 0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥ 23 = Very Severe Depression
Clinical efficacy will be measured using the Montgomery Asberg Depression Rating Scale (MADRS) | 1 year
  The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item clinician-administered scale, designed to be particularly sensitive to antidepressant treatment effects in patients with major depression. Higher scores indicate increasing depressive symptoms. Ratings can be added to form an overall score (range 0 to 50); no weights are used. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.
Clinical efficacy will be measured using the Beck Depression Inventory (BDI) | 1 year
  BDI is a self-rated depression scale. 1-10:These ups and downs are considered normal;11-16: Mild mood disturbance; 17-20: Borderline clinical depression; 21-30: Moderate depression; 31-40: Severe depression; over 40: Extreme depression.
Clinical efficacy will be measured using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 1 year
  C-SSRS is a suicidal ideation rating scale created by researchers at Columbia University to evaluate suicidality in children ages 12 and up.[1] It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent."

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No